CLINICAL TRIAL: NCT03729856
Title: Evaluation of a Novel Intervention to Promote Engagement in Physical Activity for Individuals With Whiplash Associated Disorder: a Multiple-baseline, Single Case Experimental Study
Brief Title: A Novel Intervention to Promote Engagement in Physical Activity for Individuals With Whiplash Associated Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018000349/2017/743
Record Dates: First submitted 2018-10-24; First posted 2018-11-05 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Whiplash Injuries; Sedentary Lifestyle
MeSH Terms: conditions — Whiplash Injuries; Sedentary Behavior | interventions — Methods; BaseLine dental cement

STUDY DESIGN:
Intervention Model Description: A Single Case Experimental Design (SCED) will be used to evaluate the intervention. Participants act as their own controls, and thus are exposed to both the treatment and control conditions. The study will be conducted and reported according to the Singe Case Reporting guidelines in BEhavioural Interventions (SCRIBE). A randomised, concurrent, multiple-baseline A1 (baseline control) - B (intervention)-A2 (follow-up withdrawal) design will be used to meet the methodological recommendations for SCEDs. Participants will be randomly allocated to a 5, 8 or 11 week baseline period during which they will undertake their usual activities. The baseline phase will be followed by a 16-week intervention period during which participants will participate in 12, one hour sessions with an accredited exercise physiologist. The intervention phase will be followed by a 5-week follow-up phase where participants will have no contact with the intervention personnel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- B5 week,intervention,follow-up (Experimental): Participants will undertake their usual activities for the 5 week baseline period. Participants will begin the 16 week intervention period at week 6 during which time they will participate in 12 sessions with an accredited exercise physiologist. Beginning week 22, participants will have no contact with intervention personnel during the 5 week follow-up period.
  Interventions: Behavioral: intervention; Other: B; Other: Follow-up
- B8 week,intervention,follow-up (Experimental): Participants will undertake their usual activities for the 8 week baseline period. Participants will begin the 16 week intervention period at week 9 during which time they will participate in 12 sessions with an accredited exercise physiologist. Beginning week 25, participants will have no contact with intervention personnel during the 5 week follow-up period.
  Interventions: Behavioral: intervention; Other: B; Other: Follow-up
- B11 week,intervention,follow-up (Experimental): Participants will undertake their usual activities for the 11 week baseline period. Participants will begin the 16 week intervention period at week 12 during which time they will participate in 12 sessions with an accredited exercise physiologist. Beginning week 28, participants will have no contact with intervention personnel during the 5 week follow-up period.
  Interventions: Behavioral: intervention; Other: B; Other: Follow-up

INTERVENTIONS:
Behavioral: intervention — The adapted physical activity (APA) intervention is a theory-based physical activity (PA) promotion intervention. The APA model is comprised of 4 steps: 1) pre-participation evaluation of physiological, personal and environmental factors that influence PA adoption and maintenance; 2) application of individualised, evidence based strategies associated with increased PA participation tailored to the participant's motivational readiness; 3) development of structured exercise and/or lifestyle PA program; and 4) tailored relapse prevention strategies to maintain physical activity beyond the duration of the program. The intervention will be conducted in the participant's home environment.
Other: B — Participants will undertake their usual activities during the baseline period. An extended pre-intervention time frame is needed to establish a stable control phase and enhance internal validity.
  Other Names: baseline
Other: Follow-up — Participants will have no contact with intervention personnel during the 5 week follow-up, withdrawal period. The withdrawal phase enables initial assessment of physical activity behavior change.

SUMMARY:
Approximately 50% of adults who have a whiplash injury experience ongoing pain and disability from whiplash associated disorder (WAD). Causes are multifactorial, with considerable variation. Studies evaluating interventions for this population have used group-level design and analysis and, to date, findings have been equivocal and optimal treatment remains a challenge. In addition to pain and disability, patients are frequently insufficiently active for good health, increasing their risk of preventable morbidity and mortality, and compounding the effects of WAD. The proposed study will evaluate an intervention with two novel features. Firstly, the focus is not directly on the reduction of neck pain and disability, but aims to evaluate whether evidence-based health promotion/behavior change strategies can be successfully applied to increase physical activity promotion in this population. The investigator's hypothesis is that the intervention will not only increase participation in health enhancing physical activity, but through that engagement, patients will gain increased confidence to engage in activity in the presence of neck pain, thereby reducing pain-related disability. Secondly, the Single Case Experimental Design enables individual level analysis that is not possible with typical group level designs, including identification of characteristics of responders and non-responders.

DETAILED DESCRIPTION:
Six participants will be recruited in two groups of three participants. Each group will comprise three participants who receive the same 16-week intervention (B) and 5-week follow up (maintenance), but have different lengths of the baseline period (A). The participants will be randomly allocated to one of the two groups, then subsequently randomly allocated to a baseline of either 5, 8 or 11 weeks. All participants will begin the baseline phase during the same week. Concurrent enrolment will minimize environmental influences and enhance internal validity (Kazdin, 2011). Experimental control is demonstrated by using the staggered multiple-baseline design across the participants, which controls for threats to internal validity (e.g., history, maturation) (Kazdin, 2011). The added feature of randomisation strengthens the scientific rigor of the study (Kratochwill and Levin, 2010). The design also allows for three demonstrations of the experimental effect (i.e., increased PA following the introduction of the intervention, but not before), and replication in a second group of participants (Kazdin, 2011).

During the baseline data collection period (A) participants will be encouraged to undertake their usual behaviour. Target behaviour measures (eg primary outcome measures) will be collected weekly during the baseline phase. Individual variability is addressed by repeated measurement of the target behaviour, and specifically, five data collection points within each phase is recommended to effectively evaluate a SCED intervention (Kratochwill et al., 2013).

The 16-week intervention period (B) comprises 12 one-hour intervention sessions (described below). An Accredited Exercise Physiologist (AEP) with experience in exercise prescription for individuals with a disability and behaviour change strategies associated with increasing PA will deliver the intervention. During the intervention period, the target behaviour measures will be collected fortnightly.

The intervention phase will be followed by a 5-week follow up phase where participants will have no contact with the AEP and target behaviour measures will be collected weekly. The maintenance component allows the target behavior to be monitored after the completion of the intervention, with the expectation that the target behavior will not revert to baseline levels after the intervention completion (Tate et al., 2015).

Generalisation measures (eg secondary outcome measures) will be collected at the commencement and finish of the baseline data collection period (which coincides with the intervention start point), at the end of the intervention period (which coincides with the commencement of the maintenance period), and at the end of the maintenance period; totalling 4 sampling points throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with grade II or III whiplash of at least 3 months duration;
* Individuals living in the Brisbane, Gold Coast or Northern NSW region;
* Individuals with a neck disability index score (NDI) >32% (e.g., indicative of a moderate disability);
* individuals deemed to be medically safe to participate in moderate intensity PA; and
* individuals currently not participating in structured sport or training for physical fitness; and not completing 30 minutes or more of moderate physical activity on 5 or more days per week.

Exclusion Criteria:

* presence of known or suspected serious spinal pathology;
* confirmed fracture or dislocation at time of injury (e.g., WAD Grade IV);
* nerve root compromise; and
* spinal surgery in the past 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Physical activity participation | up to 32 weeks
  Habitual physical activity measured by the ActiGraph GT9 link accelerometer. The ActiGraph is a triaxial accelerometer that measures vertical acceleration 25 times each second, and these data are integrated over a user defined or epoch, to give a number of "counts." An epoch of 1 minute will be used in this study. ActiGraph counts provide a real-time indication of the intensity of physical activity performed by an individual - the higher the counts, the greater the activity intensity. Counts will be classified as either moderate-vigorous PA (MVPA) or light/sedentary using the Freedson et al (1998) cut-point. All data collection periods will comprise a 4 day (3 week days and 1 week-end day) PA monitoring period.
Confidence in daily activities | up to 32 weeks
  A custom, single-item question to assess self-efficacy for completing daily tasks: "How confident are you in your ability to perform your daily tasks in the presence of your neck pain or disability?" with participants indicating their response on a 1 to 5 Likert scale with 1 indicating not at all confident, 3 indicating moderately confident, and 5 indicating extremely confident.
Pain interference: PROMIS- Pain interference Scale | up to 32 weeks
  Three questions of the validated PROMIS- Pain interference Scale (Amtmann et al, 2010) will be used to assess pain interference, a possible consequence of pain on relevant life aspects. These items are as follows: (a) In the past seven days, how much did pain interfere with your day to day activities?, (b) In the past seven days, how much did pain interfere with work around the home?, and (c) In the past seven days, how much did pain interfere with your ability to participate in social activities? Responses are made on a 5 point Likert-type scale with 1 = not at all; 2 = a little bit; 3 = somewhat; 4 = quite a bit; and 5 = very much.

SECONDARY OUTCOMES:
Neck disability index | up to 32 weeks
  The NDI is a valid, reliable and responsive measure of neck pain related disability (Vernon & Mior, 1991). The questionnaire has 10 items concerning pain and activities of daily living including personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation. An overall score (out of 100) will be calculated by totaling responses to 10 questions, each with 6 potential Likert-type responses (e.g., 0 indicating no disability to 5 indicating total disability), and multiplying the sum by 2 to yield a percentage.
Social support for physical activity | up to 32 weeks
  Social support will be measured using the 13-item scale developed by Sallis et al. (1987). A 5-point Likert type scale will be used to rate the frequency of support received from family and friends in the 3-months prior, with 1 indicating none, and 5 indicating very often. Social support scores will be calculated for family and friends separately by computing the sum of the items on the measure.
Decisional Balance for Physical Activity Participation | up to 32 weeks
  Decisional balance will be measured using the 16-item scale developed by Marcus et al (1992) which includes 6 items representing the avoidance of exercise (cons) and 10 items representing the positive perceptions of exercise (pros). A 5-point Likert-type scale will be used to rate how important each statement is, with 1 indicating not at all important, and 5 indicating extremely important. The average of the 10 pro items and the 6 con items will be computed. The difference in the averages (i.e., average pro score - average con score) will be taken as the decisional balance score.
Health related quality of life | up to 32 weeks
  Health related quality of life will be assessed using the Medical Outcomes Survey Short Form (SF-12). The SF-12 contains 12 questions relating to the domains physical functioning; role limitations because of physical health problems; bodily pain; general health perceptions; vitality (energy/fatigue); social functioning; role limitations because of emotional problems; and general mental health (psychological distress and psychological well-being) (Cheak-Zamora et al, 2009). Physical and mental component summary scores are computed using the 12 questions and range from 0 (lowest level of health) to 100 (highest level of health).
Numeric Pain Rating Scale | up to 32 weeks
  Participants will be asked to rate their current pain using a Numeric Pain Rating Scale (McCaffery & Beebe, 1989). Participants will be asked to select the number that best represents their pain during the previous 24-hours on a scale of 0 to 10; with 0 indicating no pain and 10 indicating worst possible pain.
Pain Catastrophizing Scale | up to 32 weeks
  The PCS is a 13-item instrument that measures the degree to which a participant has experienced specific thoughts or feelings when experiencing pain. Responses are provided on a 5-point scale with 0 indicating not at all and 4 indicating all the time. A total pain catastrophizing score may be calculated in addition to three subscales: rumination, magnification and helplessness. The total sum of responses yields a score out of 52 with higher scores indicating greater pain catastrophizing. A PCS total score >24 indicates a high level of pain catastrophizing. The PCS has been shown to have adequate internal consistency (coefficient alphas: total PCS= .87, rumination= .87, magnification= .66, and helplessness= .78) (Sullivan et al, 1995).
Pain Self-Efficacy Questionnaire | up to 32 weeks
  The Pain Self-Efficacy Questionnaire (PSEQ) is a self-administered, 10 item questionnaire survey that was developed to assess an individual's confidence to perform specific tasks in the presence of pain. Confidence in performing each of 10 activities/tasks despite current pain is rated from 0 (not at all confident) to 6 (completely confident) (Nicholas, 2007). Responses are totalled to provide a score out of 60 with higher scores reflecting stronger self-efficacy beliefs.
The Depression, Anxiety and Stress Scale short version (DASS21) | up to 32 weeks
  DASS21 is a widely used, valid and reliable self-administered tool that is designed to assess symptoms of three negative emotional states: depression, anxiety and stress (Parkitny & McAuley, 2010). The 21-item self-administered survey contains three subscales: depression, anxiety and stress. Each subscale contains 7-items. There are 4 response options for each item with 0 indicating did not apply to me at all, never and 3 indicating applied to me very much or most of the time, almost always. Scores are totalled for each subscale (Lovibond & Lovibond, 1995). Higher scores on each subscale indicate increased symptom severity.
Impact of Event Scale-Revised (IES-R) | up to 32 weeks
  The IES-R is a self-administered, 22-item survey developed to assess an individuals' subjective distress to a specific traumatic event. The IES-R comprises 3 subscales: intrusion, avoidance and hyperarousal (Weiss et al, 1999). The client is asked to report the degree of distress experienced for each item over the past 7 days. Each question has 5 response options with 0 indicating not at all and 4 indicating extremely. The scores therefore range from 0-4 for each subscale and 0-12 for the total, with higher scores indicating greater distress.
Physical activity avoidance | up to 32 weeks
  Avoidance of PA participation will be assessed using the Avoidance Subscale of the Negative Responsivity to Pain measure (Jensen et al., 2017). Participants will be asked to respond to 4 questions relating to PA avoidance. Responses are made on a 5 point Likert-type scale ranging from 0 indicating I never feel this way to 4 indicating I feel this all the time. The Negative Responsivity to Pain Measure has been shown to have excellent internal consistency and adequate test-retest reliability (Jensen et al., 2017).
Motivational readiness for change | up to 32 weeks
  Motivational readiness for change will be assessed using Marcus' Stage of Change Questionnaire (Marcus et al). This questionnaire is comprised of 4 questions relating to intention to be physically active and current activity levels. Regular physical activity in this measure is defined as 30 minutes of physical activity per day on at least 5 days of the week. Participants answer the following items using a yes or no response: I am currently physically active; I intend to become more physically active in the next 6 months; I currently engage in regular physical activity; I have been regularly physically active for the past 6 months. Yes is scored as '1' and no as '0' and a total score for the 4 questions is calculated where higher scores indicate more regular participation in physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Ritchie, PhD, Principal Investigator — The University of Queensland
Locations (1):
- The University of Queensland, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kazdin AE. Single-Case Research Designs: Methods for Clinical and Applied Settings, New York: Oxford University Press. 2011.
- [Background] Kratochwill TR, Hitchcock JH, Horner RH, et al. Single-Case Intervention Research Design Standards. Remedial and Special Education 34: 26-38, 2013.
- [Background] Kratochwill TR, Levin JR. Enhancing the scientific credibility of single-case intervention research: randomization to the rescue. Psychol Methods. 2010 Jun;15(2):124-44. doi: 10.1037/a0017736. PMID 20515235
- [Background] Tate RL, Rosenkoetter U, Wakim D, et al. (2015) The Risk of Bias in N-of-1 Trials (RoBiNT) Scale: An Expanded Manual for the Critical Appraisal of Single-Case Reports., Sydney, Australia.
- [Background] Freedson PS, Melanson E, Sirard J. Calibration of the Computer Science and Applications, Inc. accelerometer. Med Sci Sports Exerc. 1998 May;30(5):777-81. doi: 10.1097/00005768-199805000-00021. PMID 9588623
- [Background] Amtmann D, Cook KF, Jensen MP, Chen WH, Choi S, Revicki D, Cella D, Rothrock N, Keefe F, Callahan L, Lai JS. Development of a PROMIS item bank to measure pain interference. Pain. 2010 Jul;150(1):173-182. doi: 10.1016/j.pain.2010.04.025. PMID 20554116
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Sallis JF, Grossman RM, Pinski RB, Patterson TL, Nader PR. The development of scales to measure social support for diet and exercise behaviors. Prev Med. 1987 Nov;16(6):825-36. doi: 10.1016/0091-7435(87)90022-3. PMID 3432232
- [Background] Marcus BH, Rakowski W, Rossi JS. Assessing motivational readiness and decision making for exercise. Health Psychol. 1992;11(4):257-61. doi: 10.1037//0278-6133.11.4.257. PMID 1396494
- [Background] Cheak-Zamora NC, Wyrwich KW, McBride TD. Reliability and validity of the SF-12v2 in the medical expenditure panel survey. Qual Life Res. 2009 Aug;18(6):727-35. doi: 10.1007/s11136-009-9483-1. Epub 2009 May 8. PMID 19424821
- [Background] Pain: clinical manual for nursing practice Pain: clinical manual for nursing practice Margo McCaffery Alexander Beebe Mosby Yearbook UK pound17.25 0 7234 1992 2. Nurs Stand. 1994 Dec 7;9(11):55. doi: 10.7748/ns.9.11.55.s69. PMID 27527475
- [Background] Sullivan, M.J.L., S. Bishop, and J. Pivik, The Pain Catastrophizing Scale: Development and Validation. Psychological Assessment, 1995. 7: p. 524-532.
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Parkitny L, McAuley J. The Depression Anxiety Stress Scale (DASS). J Physiother. 2010;56(3):204. doi: 10.1016/s1836-9553(10)70030-8. No abstract available. PMID 20795931
- [Background] Lovibond, S. and P. Lovibond, Manual for the Depression Anxiety Stress Scales. 1995, Sydney: Psychology Foundation.
- [Background] Weiss, D., et al., The Impact of Event Scale-Revised, in Assessing Psychological Trauma and PTSD: a Practitioner's Handbook. 1999, Guilford Press: New York. p. 399-411.
- [Background] Jensen MP, Ward LC, Thorn BE, Ehde DM, Day MA. Measuring the Cognitions, Emotions, and Motivation Associated With Avoidance Behaviors in the Context of Pain: Preliminary Development of the Negative Responsivity to Pain Scales. Clin J Pain. 2017 Apr;33(4):325-334. doi: 10.1097/AJP.0000000000000407. PMID 27428549